CLINICAL TRIAL: NCT04577456
Title: Pivotal Study to Evaluate the Safety and Efficacy of the Insides™ System in the Treatment of Subjects With a Double Enterostomy and/or Enterocutaneous Fistula and Type 2 Intestinal Failure.
Brief Title: Chyme Reinfusion for Type 2 Intestinal Failure
Acronym: REINFUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Insides Company (Industry)
Collaborators: Databean (Industry); Green Lane Coordinating Centre Limited (Unknown); BioValeo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TICL-001 G190281
Record Dates: First submitted 2020-09-16; First posted 2020-10-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Intestinal Failure; Enterocutaneous Fistula; Ileostomy - Stoma; High Output Stoma
Keywords: Chyme reinfusion; Intestinal failure; TPN or PN; Parenteral nutrition; Enterocutaneous fistula; Effluent; Ileostomy - stoma; Refeeding
MeSH Terms: conditions — Intestinal Failure; Intestinal Fistula; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Global multi center prospective randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active (Experimental): Reinfusion of chyme using the Insides System for subjects with Type II intestinal failure dependent on PN
  Interventions: Device: The Insides System
- Control (No Intervention): Standard of care therapies in accordance with ASPEN and ESPEN treatment guidelines

INTERVENTIONS:
Device: The Insides System — Novel pump designed to return effluent from the ostomy bag to the distal gut
  Arms: Active

SUMMARY:
This project aims to introduce and evaluate a novel assistive prosthetic system that helps prevent and treat nutrient and fluid loss from enterocutaneous fistulas. The device system functions simply to return the output from a fistula back into the distal limb of the intestine.

DETAILED DESCRIPTION:
The development of enterocutaneous fistulas are devastating consequences of surgery or surgical diseases. They cause excessive fluid and nutrient losses from the gut resulting in severe dehydration and intestinal failure mandating invasive medical therapies to improve survival. These disorders inflict a vast burden of suffering, morbidity, and mortality on patients, while extracting enormous per-patient resources from healthcare systems. Parenteral nutrition is often required, meaning prolonged hospital stay, an attendant risk of line sepsis, venous damage and thrombosis, liver impairment, and death.

There is a pressing demand for breakthrough technologies that can restore lost fluids and nutrients to the body in patients affected by enterocutaneous fistulas in order to reverse intestinal failure, eliminate the need for parenteral nutrition, prevent dehydration and renal injury, allow safe care in the community, enable chemotherapy completion, and restore quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Able to provide written informed consent
* Dependent on parenteral nutrition (PN)
* DES/ECF with exposed afferent and efferent limbs visible on the abdominal wall
* Minimum of 2 weeks post DES/ECF creation
* Distal limb of DES/ECF opening can be intubated by a minimum 24Fr feeding tube (dilatation of orifice strictures is allowable)

Exclusion Criteria:

* Insufficient distal access channel (distal limb) for device insertion
* Bowel obstruction proximal to the DES/ECF
* Small bowel obstruction, anastomotic leak, or perforation distal to the DES/ECF (diagnostic procedure such as gastrografin test, fistulograms, or similar must be performed, if there is a distal anastomosis with integrity not previously evaluated, to ensure that the subject is eligible)
* Scheduled for DES/ECF reversal within 4 weeks of enrolment date
* Current infection with Clostridium difficile colitis
* Current infection small intestinal bacterial overgrowth (SIBO)
* Signs or symptoms of systemic infection
* Pre-existing gastrointestinal motility disorders including slow transit constipation, outlet obstruction, fecal incontinence, and gastroparesis
* Metabolic, neurogenic, or endocrine disorders known to cause colonic dysmotility, e.g., multiple sclerosis, Parkinson's disease, hypothyroidism
* Known peritoneal metastatic disease prior to DES/ECF closure (acceptable if only discovered at time of closure)
* Liver cirrhosis
* Hereditary coagulopathy, e.g., von Willebrand disease
* Severe chronic renal insufficiency prior to DES/ECF formation (eGFR<30mL/min/1.73m2)
* Active implantable medical devices such as neuromodulation and cardiac systems
* Metal stents implanted within 20cm of expected use of the controller
* Women who are pregnant or breastfeeding
* Subjects participating in an interventional clinical study within 30 days prior to randomization

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Efficacy - the proportion of subjects who achieve a 50% reduction in total caloric intake obtained from parenteral nutrition measured at 30 days post randomization compared to baseline. | 30 days post randomization
  Between group comparison of the proportion of subjects who achieve a 50% reduction in the use of parenteral nutrition

SECONDARY OUTCOMES:
Efficacy - Between group comparison of the time to reduction in the use of PN | 30 and 60 days
  Between group comparison of the time to reduction of parenteral nutrition measured in days
Efficacy - Between group comparison of the time to discontinuation in the use of PN | 30 and 60 days
  Between group comparison of the time to discontinuation in the use of PN
Efficacy - Between group comparison of the time to reduction in the use of other parentral support fluids | 30 and 60 days
  Between group comparison of the time to reduction in the use of other parenteral support fluids
Safety - Between group comparison of the incidence of serious adverse events | 30 and 60 days
  Between group comparison of the incidence of serious adverse events such as dehydration, metabolic disarray, failure to complete prescribed chemotherapy, IV line complications, fistula complications, device related effects
Efficacy - Between group comparison of the time to ostomy closure | 30 and 60 days
  Between group comparison of the time to surgery for ostomy closure measured in days
Safety - Between group comparison of medication use to control fluid loss due to high output enterostomies | 30 and 60 days
  Between group comparison of the use of proton pump inhibitors, anti motility agents, histamine receptor antagonists, a2 receptor antagonists, and somatostatins.
Safety - Between group comparison of nutritional failure measured by the nutritional risk index (NRI) | 30 and 60 days
  Between group comparison of the nutritional risk index (NRI). Nutritional failure risk will be categorized as severe (NRI<83.5), moderate (NRI 83.5 - 97.5) and low (NRI>97.5).
Safety - Between group comparison of peristomal skin complications | 30 and 60 days
  Between group comparison of peristomal skin complications measured by the discoloration, erosion, tissue overgrowth (DET) score as mild, moderate or severe
Healthcare Utilization - Between group comparison of length of stay for index hospitalization | up to 30 days
  Between group comparison of length of stay for index hospitalization measured from the day of randomization to discharge
Healthcare Utilization - Between group comparison of all cause hospitalizations | 30 and 60 days
  Between group comparison of all cause hospitalizations measured by the total number of discreet hospitalizations >24 hours in duration
Healthcare Utilization - Between group comparison of hospitalizations due to dehydration | 30 and 60 days
  Between group comparison of hospital admissions >24 hours duration where the primary reason for admission is dehydration
Device performance - The overall incidence of device related adverse effects | 30 and 60 days
  The overall incidence of device related adverse effects reported in subjects randomized to the device. Effects may include effluent cycling time, device wear, device failure.
Quality of Life - Between group comparison of quality of life indices as measured by the EuroQol 5D | 30 and 60 days
  Between group comparison of quality of life as measured by the EQ-5D-3L - a survey of the following five health dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and a health thermometer where 0= the worst health you can imagine and 100= the best health you can imagine.
Quality of Life - Between group comparison of quality of life indices as measured by the Stoma QoL Questionnaire | 30 and 60 days
  Stoma QoL - This questionnaire consists of 20 questions. An example of a question could be: "I worry that the pouch will loosen." All the questions must be answered on a 4-point scale. The options for answering each question are:
  1. Always
  2. Sometimes
  3. Rarely
  4. Not at all
Quality of Life - Between group comparison of quality of life indices as measured by the Beck Depression Inventory | 30 and 60 days
  Beck Depression Inventory - a 21 question survey where each question has 4 possible answers scored 0-3. The total score is summed to give an overall level of depression
  1-10____________________These ups and downs are considered normal 11-16___________________ Mild mood disturbance 17-20___________________Borderline clinical depression 21-30___________________Moderate depression 31-40___________________Severe depression over 40__________________Extreme depression

CONTACTS AND LOCATIONS:
Overall Officials: Dermot Burke, MD, Principal Investigator — St. James Hospital, Leeds, UK
Locations (11):
- United States (4):
  - Shands Hospital, Gainesville, Florida
  - University Miami Hospital and Clinics, Miami, Florida
  - University Illinois, Chicago, Illinois
  - University Nebraska, Lincoln, Nebraska
- United Kingdom (7):
  - Royal Devon and Exeter Hospital, Exeter
  - St James's Hospital, Leeds
  - St Mark's Hospital, London
  - Salford Royal Hospital, Manchester
  - Royal Victoria Hospital, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No